CLINICAL TRIAL: NCT00090090
Title: A Multi-Center, Open-Label, Non-Randomized Phase II Study of Elsamitrucin (SPI 28090) In Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Elsamitrucin (SPI 28090) for Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELSA 2004-001
Record Dates: First submitted 2004-08-24; First posted 2004-08-25 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Mantle Cell Lymphoma; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — elsamicin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Elsamitrucin

SUMMARY:
To determine the safety and efficacy of elsamitrucin in patients with relapsed or refractory non-Hodgkin's lymphoma (NHL). To determine if elsamitrucin is efficacious in a particular pathologic NHL subtype(s).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or Refractory mantle cell lymphoma and/or CLL/SLL except Burkitt's, Burkitt's like or HIV-associated lymphoma
* at least one prior cytotoxic chemotherapy regimens
* measurable disease
* adequate bone marrow, liver and kidney function
* ECOG PS 0-2

Exclusion Criteria:

* prior treatment with elsamitrucin
* prior chemo, antibody or radiotherapy for NHL within 28 days prior to start to treatment
* HIV positive or known AIDS syndrome
* uncontrolled medical disease or psychiatric condition/s

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114
Dates: Start 2004-04; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Alta Bates Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - USC Norris Cancer Center, Los Angeles, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - North Valley Hematology Oncology Medical Group, Mission Hills, California
  - Cancer and Blood Institute Medical Group, Rancho Mirage, California
  - North Shores University Hospital, Manhasset, New York

REFERENCES:
- [Background] Allen SL, Schacter LP, Lichtman SM, Bukowski R, Fusco D, Hensley M, O'Dwyer P, Mittelman A, Rosenbloom B, Huybensz S. Phase II study of elsamitrucin (BMY-28090) for the treatment of patients with refractory/relapsed non-Hodgkin's lymphoma. Invest New Drugs. 1996;14(2):213-7. doi: 10.1007/BF00210793. PMID 8913843